CLINICAL TRIAL: NCT07368114
Title: Validity of Ozonated Olive Oil Gel Versus Injectable Bone Graft on Osseointegration of Immediate Dental Implants
Brief Title: Validity of Ozonated Olive Oil Gel Versus Injectable Bone Graft
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 738/2023
Record Dates: First submitted 2026-01-08; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2023-10

CONDITIONS: Dental; Implant Osseointegration; Ozone Therapy; Bone Graft
Keywords: Osseointegration; Dental Implants; Ozonated Olive Oil Gel; Injectable Bone Graft
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 16 immediate implants will be placed in the mandibular premolar region, divided randomly into two groups: Group 1 (control) will use injectable bone graft for 8 implants, while Group 2 (study) will use ozonated olive oil gel as graft material for the other 8 implants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Control Group) (Active Comparator): 8 implants were inserted immediately after teeth extraction with grafting of injectable β-tricalcium phosphate (β-TCP) bone graft around the implant.
  Interventions: Procedure: Immediate implant placement; Biological: β-tricalcium phosphate Injectable Bone Graft
- Group II (Study Group) (Experimental): 8 implants were inserted immediately after teeth extraction with grafting of ozonated olive oil gel around the implant.
  Interventions: Procedure: Immediate implant placement; Biological: Ozonated olive oil gel

INTERVENTIONS:
Procedure: Immediate implant placement — Placement of a dental implant immediately after tooth extraction in the mandibular premolar region following standard surgical protocol.
Biological: β-tricalcium phosphate Injectable Bone Graft — Immediate implant placement in the mandibular premolar region with application of injectable bone graft material to the peri-implant defect.
  Other Names: Group I; Control Group
  Arms: Group I (Control Group)
Biological: Ozonated olive oil gel — Immediate implant placement in the mandibular premolar region with application of ozonated olive oil gel to the peri-implant defect.
  Other Names: Group II; Study Group
  Arms: Group II (Study Group)

SUMMARY:
Many of studies have been performed to improve osseointegration and bone density around implants by modifying the implant by adding bone graft or substitute material that increase success of implant. The aim of this study is to evaluate clinically and radiographically the efficacy of injectable bone graft versus ozonated olive oil gel to promote bone formation and improve outcomes in immediate implant cases. 16 immediate implants will be placed in mandibular premolar region the study will be devided equally and randomlly into two groups , Group 1: it will be 8 immediate implants represent the control group were the implants will be placed with injectable bone graft , Group 2: will be 8 immediate implant represent the study group were the implants will be placed with ozonated olive oil gel be used as a graft material . The implant stability will be assessed clinically using Ostell , and the bone density will be assed radiographically .

ELIGIBILITY:
Inclusion criteria:

* Adults aged between 20 and 60 years.
* Adults of both genders.
* Patients who are medically healthy and without systemic conditions that could contraindicate implant placement.
* Patients requiring extraction of a single unrestorable mandibular premolar indicated for immediate implant placement.
* Presence of sufficient apical and peripheral bone to achieve primary implant stability (minimum 3-5 mm of bone beyond the socket apex and overall socket length ≥ 10 mm).

Exclusion criteria:

* Pregnant and lactating women's
* Heavy smoking (>10 cigarettes/day)
* Severe parafunctional habits (e.g., uncontrolled bruxism).
* Periapical infections or lesions.
* Gingival and periodontal diseases.
* Inability or unwillingness to attend scheduled follow-up visits.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Implant Stability (ISQ) | Baseline, and 6 months postoperatively
  Osstell enables precise and objective monitoring of osseointegration and implant stability through non-invasive measurements. A cable-connected probe requires a smart peg to be securely attached to the implant. When using the device, it should be held at a right angle to the implant, with a maximum deviation of 45 degrees and a distance of 0.6-2.5 mm from the test surface. The implant stability is measured using the ISQ scale, ranging from 1 to 100, where values above 70 indicate strong stability, 60-69 indicate medium stability, and lower values suggest lower stability. Measurements are taken immediately postoperatively and reassessed after 6 months for final stability confirmation.
Bone density | Baseline, 3 and 6 months postoperatively
  Direct paralleling digital periapical radiographs were obtained using the KaVo Scan eXam™ One system and the Rinn extension cone paralleling device. The KaVo system employs a thin, flexible, wireless phosphorescent imaging plate, and the imaging plate size 2 has a specific active surface area and resolution. A long cone was attached to the x-ray tube, and fixed exposure parameters were applied throughout the study. Radiographic assessments occurred immediately post-operative and after 3 and 6 months. Image analysis utilized IDRISI Kilimanjaro software for restoration, enhancement, and densitometric measurements. This software uniquely monitored changes in bone density in two zones: the osseointegration zone near the implant border and the surrounding bone interface.

SECONDARY OUTCOMES:
Visual Analogue Scale of Pain (VAS) | Days 1, 3, and 7 postoperatively
  The Visual Analog Scale (VAS) is a widely utilized instrument for quantifying pain intensity in clinical settings. It features a 10-centimeter horizontal line marked at both ends to represent the range of possible pain experiences, where one end is typically labeled "no pain" and the opposite end may carry descriptors such as "unimaginably unspeakable pain." Patients are instructed to indicate their pain level by placing a mark on the line that corresponds to their current pain experience. The measurement in centimeters from the "no pain" endpoint to the patient's designated point provides a straightforward numerical representation of pain severity. This method is favored for its simplicity and its ability to yield quantifiable data, facilitating better pain assessment and management in various medical contexts.
Visual Scale of Edema | Days 1, 3, and 7 postoperatively
  Facial edema was assessed using a clinical grading scale based on visual inspection and palpation, classifying it into four severity categories: No Edema (normal contours and symmetry), Low-grade Edema (mild swelling without functional limitations), Intermediate-grade Edema (moderate swelling with visible asymmetry and slight discomfort), and High-grade Edema (pronounced swelling with evident asymmetry and significant functional interference).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Said Hamed, Professor, Study Chair — Professor of Oral and Maxillofacial Surgery, Faculty of Dentistry - Suez Canal University; Shimaa Abdallah Metawea, B.D.S, Principal Investigator — Dentist at Ministry of Health and Population; Ahmed Mohamed El Rawdy, Professor, Study Director — Professor of Oral and Maxillofacial Radiology, Faculty of Dentistry - Suez Canal University; Ahmed Abd elmohsen Younis, Assistant. Professor, Study Director — Assistant. Professor of Oral and Maxillofacial Surgery, Faculty of Dentistry - Suez Canal University
Locations (1):
- Suez Canal University, Faculty of Dentistry, Ismailia, Egypt

REFERENCES:
- [Background] Botticelli D, Renzi A, Lindhe J, Berglundh T. Implants in fresh extraction sockets: a prospective 5-year follow-up clinical study. Clin Oral Implants Res. 2008 Dec;19(12):1226-32. doi: 10.1111/j.1600-0501.2008.01620.x. PMID 19040437
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- [Background] Abas, M., Ghanem, W., El Desouky, G., El Gerby, Y. (2021). 'Clinical and Radiographic Evaluation of Immediate Implant with Bone Graft (Hyprooss)', Dental Science Updates, 2(1), pp. 17-25.
- [Result] Barone S, Zaffino P, Salviati M, Destito M, Antonelli A, Bennardo F, Cevidanes L, Spadea MF, Giudice A. Automated pipeline for linear and volumetric assessment of facial swelling after third molar surgery. BMC Oral Health. 2024 Nov 19;24(1):1404. doi: 10.1186/s12903-024-05193-7. PMID 39563399